CLINICAL TRIAL: NCT05859165
Title: Clinical Efficacy and Safety of Diabetes-Specific Formula (Nutren Diabetes) for Nutritional Support in Diabetic Patients With Dysphagia
Brief Title: To Evaluate Clinical Efficacy and Safety of Diabetes-Specific Formula (Nutren Diabetes)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: Nestle Health Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22.01.CN.NHS
Record Dates: First submitted 2023-05-04; First posted 2023-05-15 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutren Diabetes group (Experimental): Product Replacement phase: 1-5 days, tube-feeding, 25kcal/kg/day Formal intervention phase:7 days, tube-feeding, 25kcal/kg/day
  Interventions: Dietary Supplement: Nutren Diabetes
- Fresubin Diabetes group (Active Comparator): Product Replacement phase: 1-5 days, tube-feeding, 25kcal/kg/day Formal intervention phase:7 days, tube-feeding, 25kcal/kg/day
  Interventions: Dietary Supplement: Fresubin Diabetes

INTERVENTIONS:
Dietary Supplement: Nutren Diabetes — Product replace phase: 1-5 days, tube feeding, 25kcal/kg/day Formal intervention phase:7 days, tube feeding, 25kcal/kg/day
  Arms: Nutren Diabetes group
Dietary Supplement: Fresubin Diabetes — Product replace phase: 1-5 days, tube feeding, 25kcal/kg/day Formal intervention phase:7 days, tube feeding, 25kcal/kg/day
  Arms: Fresubin Diabetes group

SUMMARY:
This study has a parallel, non-inferiority design, comparing the 24h AUC of Nutren Diabetes group with Fresubin Diabetes group at 2-4 days since the start of formal intervention.

DETAILED DESCRIPTION:
This is a randomized, active-control, open labelled study in which either Nutren Diabetes or Fresubin Diabetes will be given to patients with diabetes for around 9 days.

24h AUC, TIR, TBR, prealbumin albumin etc. will be evaluated. And also safety-related laboratory parameters, numbers, severity, outcome of AEs will be evaluated too.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-90 years old (inclusive);
* The subjects' blood glucose related indicators meet any of the following conditions:

Diagnosis of diabetes, and recent stable blood glucose control (refer to Guidelines for the Prevention and Treatment of Type 2 Diabetes Mellitus in China (2020) for the diagnosis of diabetes); Fasting blood glucose ≥ 7.0mmol/L or random blood glucose ≥ 11.1mmol/L (at least 2 consecutive tests); Blood glucose>7.8mmol/L (at least 3 consecutive tests, with at least 2 non same day results).

* Glycosylated hemoglobin (HbA1c) <10.0%;
* Inability to feed orally;
* It is estimated that tube feeding would be required for more than 9 days;
* Patients or their guardians (or authorized personnel) have fully understood the study procedures of this trial and are willing to sign the informed consent form (ICF).

Exclusion Criteria:

* Subjects with congenital metabolism disorder or allergy to any ingredient in the product (such as whey protein, milk protein concentrate, soybean lecithin); those with congenital intolerance to fructose;
* Patients who are not suitable for enteral nutrition, such as those with active gastrointestinal (GI) hemorrhage, intestinal ischemia, paralytic/mechanical ileus, decreased GI tension, stress ulcer, as well as severe abdominal distension, diarrhea and other digestive and absorptive dysfunction. If the above situation exists, but the researchers believe that enteral nutrition is still applicable, screening can be conducted;
* Subjects with severe local broken skin which affects the use of continuous glucose monitoring (CGM) system;
* Subjects who have concurrent severe malnutrition (body mass index [BMI] <15), severe hypertriglyceridemia (triglyceride≥5.6 mmol/L), severe hypoproteinemia (albumin<20 g/L), severe immunosuppression (neutrophils<1500/mm3 or lymphocytes<500/mm3), severe anemia (hemoglobin<60 g/L), severe infection, high fever and other stress conditions;;
* Subjects with fasting C-peptide < 100 pmol/L (0.3 ng/mL);
* Patients with active malignant tumor (except for glioma, meningioma) or in the period of radiochemotherapy;
* Patients with severe cardiac failure (New York Heart Association [NYHA] Class IV); those with severe liver or renal impaired function (glomerular filtration rate < 30 mL/min/1.73 m2, or levels of transaminases or transpeptidases more than 3 times the upper limit of normal); or those with conditions such as active hyperthyroidism, treatment-resistant hypothyroidism;
* Subjects with one of the following conditions: hemodynamic instability, life-threatening multiple injuries, as well as severe acidosis, shock, sepsis;
* Recent (within 3 months) acute complications of diabetes, such as diabetic ketoacidosis, hyperosmolar hyperglycemic syndrome;
* Subjects who have used systemic glucocorticoid therapy within 2 weeks prior to screening or are expected to use during the study, If the screening requires the use of physiological replacement doses of glucocorticoids for other diseases prior to screening, and the researcher evaluates that the glucocorticoid dose can remain stable during the study period, the subjects can be screened;
* Women who are pregnant or plan to become pregnant or are breastfeeding;
* Life expectancy ≤ 30 days;
* Participated in other interventional clinical trials within 4 weeks prior to screening, including those involved in drugs, nutritional preparations, medical devices, etc.;
* Other cases not eligible for this study in the investigator's opinion, such as inflammatory bowel disease (Crohn's disease or ulcerative colitis), acute pancreatitis, unstable vital signs, and if it does, the reasons for ineligibility should be recorded.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-03-18 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
24h AUC of Nutren Diabetes group with Fresubin Diabetes group | 2-4 days since the start of formal intervention
  mean area under the blood glucose concentration-time curve from time 0 to 24h (24h AUC)

SECONDARY OUTCOMES:
Coefficient of variation of blood glucose | Day 2 upon formal intervention
  CV data from CGM
Time in range | Day 2 - 4 upon formal intervention
  TIR from CGM
Time above range | Day 2 - 4 upon formal intervention
  TAR from CGM
Time below range | Day 2 - 4 upon formal intervention
  TBR from CGM
Mean amplitude of glycemic excursion | Day 2 - 4 upon formal intervention
  MAGE from CGM
Peak blood glucose | Day 4 upon formal intervention
  Peak blood from CGM
Fasting plasma glucose | Day 7 upon formal intervention
  FPG from laboratory test
Prealbumin | Day 7 upon formal intervention
  Prealbumin from laboratory test
Albumin | Day 7 upon formal intervention
  Albumin from laboratory test

CONTACTS AND LOCATIONS:
Overall Officials: Wei Chen, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No